CLINICAL TRIAL: NCT00724308
Title: Telephone Care Coordination for Smokers in Mental Health Clinics
Brief Title: Telephone Care Coordination for Smokers in VA Mental Health Clinics
Acronym: TeleQuit MH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: SDP 07-034
Record Dates: First submitted 2008-07-23; First posted 2008-07-29 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2020-11-17 (Actual); Status verified 2020-10

CONDITIONS: Smoking
Keywords: Smoking; Smoking Cessation; Tobacco; Mental Health
MeSH Terms: conditions — Smoking; Smoking Cessation; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Experimental): The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from TeleQuit MH study counselors; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
  Interventions: Other: Telephone Care Coordination
- Arm 2 (Experimental): The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from the patient's state smoking cessation "Quitline"; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
  Interventions: Other: Telephone Care Coordination with state Quitline

INTERVENTIONS:
Other: Telephone Care Coordination — The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from TeleQuit MH study counselors; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
  Arms: Arm 1
Other: Telephone Care Coordination with state Quitline — The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from the patient's state "Quitline"; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
  Arms: Arm 2

SUMMARY:
The purpose of this study is to evaluate whether a smoking cessation telephone care coordination program is effective and feasible in VA Mental Health Clinics.

DETAILED DESCRIPTION:
Smoking is the leading preventable cause of death in the United States and is a particular problem among VA users and among persons with a diagnosed mental illness. The prevalence of smoking among VA mental health patients has remained high, in part because smoking cessation treatment rates have remained low. Telephone-based counseling represents the most feasible approach to increasing smoking cessation treatment among VA patients. The approach used in this study has been used very effectively in a primary care-based population that includes a large percentage of mental health patients. This project would target the program specifically at patients seen in VA Mental Health Clinics.

ELIGIBILITY:
Inclusion Criteria:

* Smokers who are referred from Mental Health Clinics in VA VISNs 1 and 3.
* Patients must have access to a telephone and a regular mailing address.

Exclusion Criteria:

* No access to a telephone
* no mailing address
* not receiving care from a VISN 1 or VISN 3 Mental Health provider

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 577 (Actual)
Dates: Start 2009-11; Primary Completion 2012-10 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott E Sherman, MD MPH, Principal Investigator — Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY
Locations (1):
- Manhattan Campus of the VA NY Harbor Healthcare System, New York, NY, New York, New York, United States

REFERENCES:
- [Result] Rogers E, Fernandez S, Gillespie C, Smelson D, Hagedorn HJ, Elbel B, Kalman D, Axtmayer A, Kurowski K, Sherman SE. Telephone care coordination for smokers in VA mental health clinics: protocol for a hybrid type-2 effectiveness-implementation trial. Addict Sci Clin Pract. 2013 Mar 15;8(1):7. doi: 10.1186/1940-0640-8-7. PMID 23497630
- [Result] Rogers ES, Gillespie C, Zabar S, Sherman SE. Using standardized patients to train telephone counselors for a clinical trial. BMC Res Notes. 2014 Jun 5;7:341. doi: 10.1186/1756-0500-7-341. PMID 24903609
- [Derived] Swong S, Nicholson A, Smelson D, Rogers ES, El-Shahawy O, Sherman SE. The effectiveness of a telephone smoking cessation program in mental health clinic patients by level of mental well-being and functioning: a secondary data analysis of a randomized clinical trial. BMC Public Health. 2023 Nov 7;23(1):2190. doi: 10.1186/s12889-023-16975-z. PMID 37936218
- [Derived] Swong S, Nicholson A, Smelson D, Rogers ES, El-Shahawy O, Sherman SE. The Effectiveness of a Telephone Smoking Cessation Program in Mental Health Clinic Patients by Level of Mental Well-Being and Functioning: A Secondary Data Analysis of a Randomized Clinical Trial. Res Sq [Preprint]. 2023 Aug 24:rs.3.rs-3179446. doi: 10.21203/rs.3.rs-3179446/v1. PMID 37674733
- [Derived] Rogers ES, Smelson DA, Gillespie CC, Elbel B, Poole S, Hagedorn HJ, Kalman D, Krebs P, Fang Y, Wang B, Sherman SE. Telephone Smoking-Cessation Counseling for Smokers in Mental Health Clinics: A Patient-Randomized Controlled Trial. Am J Prev Med. 2016 Apr;50(4):518-527. doi: 10.1016/j.amepre.2015.10.004. Epub 2015 Dec 17. PMID 26711163

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm 1 - VA Counselling: Telephone Care Coordination with VA counselors: The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from a VA counselor; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
- Arm 2 - Quitline Counseling: Telephone Care Coordination with state Quitline: The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) warm transfer to state "Quitline" for cessation counseling; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
Period: Overall Study
Arm/Group | Arm 1 - VA Counselling | Arm 2 - Quitline Counseling
Started | 270 | 307
Completed | 190 | 210
Not Completed | 80 | 97

BASELINE CHARACTERISTICS:
Groups:
- Arm 1 - VA Counseling: Telephone Care Coordination with VA counselors: The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from a VA counselor; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
- Total: Total of all reporting groups
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling | Total
Number analyzed (Participants) | 270 | 307 | 577
Age, Continuous [Mean (Standard Deviation); unit: years] | 54 (12) | 54 (12) | 54 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 21 | 43
  Male | 248 | 286 | 534
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 3 | 6
  Asian | 1 | 3 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 92 | 114 | 206
  White | 151 | 169 | 320
  More than one race | 22 | 15 | 37
  Unknown or Not Reported | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Long-term Smoking Abstinence (30-day Point Prevalence Abstinence)
Time Frame: 6 months after enrollment
Measure: Number; unit: participants
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling
Number analyzed (Participants) | 190 | 210
participants | 49 | 38

2. Secondary Outcome: 30-day Point Prevalence Abstinence Rate at 2-months (i.e., End of Treatment)
Time Frame: 2 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling
Number analyzed (Participants) | 211 | 232
Participants | 38 | 32

3. Secondary Outcome: Quit Attempt Rate
Time Frame: 2 and 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling
Number analyzed (Participants) | 270 | 307
Participants
  2-months | 137 | 169
  6-months | 156 | 165

4. Secondary Outcome: Rate of Use of Smoking Cessation Medications (i.e., Treatment Rate)
Time Frame: 2 and 6 months after enrollment
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling
Number analyzed (Participants) | 270 | 307
Participants
  NRT - 6 months | 124 | 157
  Bupropion - 6 months | 243 | 269

5. Secondary Outcome: VA Site-level Performance Rates on the VA Tobacco Performance Measures
Time Frame: Quarterly after study implementation
Population: Participants could receive more than one type of treatment, therefore counts do not necessarily sum to the total number of participants.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1 - VA Counseling | Arm 2 - Quitline Counseling
Number analyzed (Participants) | 270 | 307
Participants
  Counselling - 6 months : NY Harbor HCS: number analyzed (Participants) | 153 | 155
  Counselling - 6 months : NY Harbor HCS | 75 | 35
  Counselling - 6 months : Bedford: number analyzed (Participants) | 3 | 8
  Counselling - 6 months : Bedford | 0 | 3
  Counselling - 6 months : NJ HCS: number analyzed (Participants) | 39 | 50
  Counselling - 6 months : NJ HCS | 22 | 20
  Counselling - 6 months : Bronx: number analyzed (Participants) | 32 | 45
  Counselling - 6 months : Bronx | 18 | 14
  Counselling - 6 months : Providence: number analyzed (Participants) | 15 | 17
  Counselling - 6 months : Providence | 3 | 8
  Counselling - 6 months : White River Junction: number analyzed (Participants) | 28 | 32
  Counselling - 6 months : White River Junction | 10 | 8
  NRT - 6 months : NY Harbor HCS: number analyzed (Participants) | 153 | 155
  NRT - 6 months : NY Harbor HCS | 83 | 78
  NRT - 6 months : Bedford: number analyzed (Participants) | 3 | 8
  NRT - 6 months : Bedford | 0 | 3
  NRT - 6 months : NJ HCS: number analyzed (Participants) | 39 | 50
  NRT - 6 months : NJ HCS | 20 | 29
  NRT - 6 months : Bronx: number analyzed (Participants) | 32 | 45
  NRT - 6 months : Bronx | 19 | 18
  NRT - 6 months : Providence: number analyzed (Participants) | 15 | 17
  NRT - 6 months : Providence | 7 | 7
  NRT - 6 months : White River Junction: number analyzed (Participants) | 28 | 32
  NRT - 6 months : White River Junction | 17 | 15
  Bupropion - 6 months : NY Harbor HCS: number analyzed (Participants) | 153 | 155
  Bupropion - 6 months : NY Harbor HCS | 16 | 18
  Bupropion - 6 months : Bedford: number analyzed (Participants) | 3 | 8
  Bupropion - 6 months : Bedford | 0 | 1
  Bupropion - 6 months : NJ HCS: number analyzed (Participants) | 39 | 50
  Bupropion - 6 months : NJ HCS | 6 | 7
  Bupropion - 6 months : Bronx: number analyzed (Participants) | 32 | 45
  Bupropion - 6 months : Bronx | 4 | 6
  Bupropion - 6 months : Providence: number analyzed (Participants) | 15 | 17
  Bupropion - 6 months : Providence | 0 | 1
  Bupropion - 6 months : White River Junction: number analyzed (Participants) | 28 | 32
  Bupropion - 6 months : White River Junction | 1 | 5

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Arm 1: Telephone Care Coordination with VA counselors: The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) proactive multi-call counseling from a VA counselor; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
- Arm 2: Telephone Care Coordination with state Quitline: The telephone care coordination program involves the following steps: (1) brief counseling and referral from a mental health provider; (2) prescribing and mailing of smoking cessation medications; (3) warm transfer to state "Quitline" for cessation counseling; and (4) follow-up at 2 and 6 months to check the patient's smoking status.
Arm/Group | Arm 1 | Arm 2
Serious Adverse Events (participants affected / at risk) | 0/270 | 0/307
Other Adverse Events (participants affected / at risk) | 0/270 | 0/307

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No